CLINICAL TRIAL: NCT01542710
Title: Bimatoprost/Timolol Versus Travoprost/Timolol Fixed Combinations in an Egyptian Population: A Hospital-Based Prospective Randomized Study
Brief Title: Bimatoprost/Timolol Versus Travoprost/Timolol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tamer A Macky, Assistant Professor, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fixed Glaucoma Medications; GFDU-2011; GANDUO-2011 (Other: Cairo University)
Record Dates: First submitted 2012-02-06; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2011-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Ganfort; Bimatoprost; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glaucoma fixed Combination Medications (Experimental)
  Interventions: Drug: Ganfort; Drug: Duotrav

INTERVENTIONS:
Drug: Ganfort — Bimatoprost/Timolol fixed combination
  Other Names: Bimatoprost/Timolol vs Travoprost/Timolol fixed combination
Drug: Duotrav — Fixed combination of Travoprost and Timolol

SUMMARY:
The purpose of this study is to compare 2 fixed combination medications in intraocular pressure lowering.

DETAILED DESCRIPTION:
PURPOSE: To compare the efficacy of bimatoprost/timolol (BTFC) or travoprost/timolol (TTFC) fixed combinations on intraocular pressure (IOP) reduction in an Egyptian population.

METHODS: Patients with primary open angle glaucoma (POAG) were randomized to receive either BTFC or TTFC. IOPs were measured at baseline, 2 weeks, and 1, 2, 4, and 6 months. The primary outcome measures were the mean change in IOP from baseline

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma

Exclusion Criteria:

* No other ocular diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of drop of intraocular pressures from baseline. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tamer A Macky, MD FRCS, Principal Investigator — Cairo University
Locations (1):
- Kasr El Aini Hospital, Cairo, Egypt